CLINICAL TRIAL: NCT02759523
Title: Neural Mechanisms Underlying Children's Responses to Food Portion Size and Energy Density
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Collaborators: Social Science Research Institute (Unknown)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Director, Metabolic Kitchen & Children's Eating Behavior Lab, Penn State University
Other Study IDs: FoodBehavior01
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Pediatric Obesity
Keywords: Magnetic Resonance Imaging; Portion Size; Energy Intake
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Increased portion sizes of foods high in energy density (calories per gram of food) have been implicated in the obesity epidemic. Numerous studies show that children and adults eat more from larger portions of food than they do from smaller portions, a response known as the portion size effect. Despite the robust and consistent nature of these findings, the mechanisms underlying the portion size effect are not known. The long-term goal of this research is to identify the neural mechanisms involved in the portion size effect so that this information can be used to develop effective weight-management strategies. Differences in neural response to food cues, as demonstrated by functional magnetic resonance imaging (fMRI), can help clarify the factors that determine susceptibility to large portions. The goal of this study is to identify brain regions activated in response to portion size and energy density and relate these neural responses to laboratory eating behaviors in children.

The investigators hypothesize that high relative to low energy density food images will be associated with increased activation in regions of the brain involved in reward- and sensory- processing and that large relative to small portion size food images will be associated with increased activation in regions of the brain involved in cognitive control. In addition, the investigators hypothesize that these brain responses will influence the relationship between portion size served and energy intake at laboratory meals.

DETAILED DESCRIPTION:
What this study will add to the literature: The response to food images that vary by portion size using fMRI has not been previously reported. Furthermore, how the brain response to food portion size and energy density is related to energy intake has not been previously reported. The goal of this study is to identify brain regions activated in response to portion size and energy density and relate these neural responses to laboratory eating behaviors in children.

ELIGIBILITY:
Inclusion Criteria:

* Right-handedness
* English as native language
* Reading at /above grade level
* Not claustrophobic
* Generally healthy

Exclusion Criteria:

* Left-handedness
* Metal in or on the body that cannot be removed
* Claustrophobic
* Medication usage that could alter brain activity
* Medical disorder that may impact comfort in scanner
* Food allergies

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between the ages of 7-10 years old and their parents
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
fMRI blood oxygen level dependent (BOLD) response to food portion size and energy density | Collected at fMRI scan (1 of 1) at week 5
  Whole-brain response to food images that varied at 2 levels of portion size and 2 levels of energy density
Energy intake | Collected at week 1, 2, 3, and 4
  Energy intake (kcal and grams) of foods consumed ad libitum at each laboratory test-meal in response to 4 conditions of portion sizes (100% reference, 133%, 167%, 200%).

SECONDARY OUTCOMES:
Region of Interest (ROI)-response to food portion size and energy density | Collected at fMRI scan (1 of 1) at week 5
  Response in selected brain regions of interest to food images varied at 2 levels of portion size and 2 levels of energy density

OTHER OUTCOMES:
Appetitive traits | Collected at week 1 (Baseline)
  Parent-reported questionnaire of habitual eating styles in children
Body composition a/o weight status | Collected at week 1 (Baseline)
  Height, weight and body fat percentage were measured. Body mass index (BMI), BMI z score, fat-mass index and fat-free-mass index will be calculated.
Liking of foods | Collected at week 5
  Ratings of how much child likes food presented on a computerized visual analog scale
Wanting of foods | Collected at week 5
  Ratings of how much child wants food presented on a computerized visual analog scale
Loss of control eating | Collected at week 1 (Baseline)
  Loss of control when eating is frequently reported in middle childhood. Loss of control when eating was assessed via interview-style questionnaire to determine pre-clinical binge-like eating behaviors that may influence the primary outcome of energy intake at the 4 conditions of test-meals.
Parental feeding strategies | Collected at week 1 (Baseline)
  Parent-reported measures of feeding practices

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Keller, PhD, Principal Investigator — The Pennsylvania State University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] English L, Lasschuijt M, Keller KL. Mechanisms of the portion size effect. What is known and where do we go from here? Appetite. 2015 May;88:39-49. doi: 10.1016/j.appet.2014.11.004. Epub 2014 Nov 11. PMID 25447010
- [Result] Fearnbach SN, English LK, Lasschuijt M, Wilson SJ, Savage JS, Fisher JO, Rolls BJ, Keller KL. Brain response to images of food varying in energy density is associated with body composition in 7- to 10-year-old children: Results of an exploratory study. Physiol Behav. 2016 Aug 1;162:3-9. doi: 10.1016/j.physbeh.2016.03.007. Epub 2016 Mar 10. PMID 26973134
- [Derived] Diktas HE, Keller KL, Roe LS, Rolls BJ. Children's Portion Selection Is Predicted by Food Liking and Is Related to Intake in Response to Increased Portions. J Nutr. 2022 Oct 6;152(10):2287-2296. doi: 10.1093/jn/nxac162. PMID 35883226
- [Derived] Keller KL, English LK, Fearnbach SN, Lasschuijt M, Anderson K, Bermudez M, Fisher JO, Rolls BJ, Wilson SJ. Brain response to food cues varying in portion size is associated with individual differences in the portion size effect in children. Appetite. 2018 Jun 1;125:139-151. doi: 10.1016/j.appet.2018.01.027. Epub 2018 Feb 2. PMID 29408590